CLINICAL TRIAL: NCT05554107
Title: The Effect of Physical Activity on Postural Orthostatic Tachycardia Syndrome
Acronym: POTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: POTS-phys
Record Dates: First submitted 2022-09-21; First posted 2022-09-26 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: POTS - Postural Orthostatic Tachycardia Syndrome
Keywords: Exercise; POTS; Training programme; Treatment; Orthostatic intolerance
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome; Motor Activity; Orthostatic Intolerance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A - Supervised exercise first (Active Comparator): All POTS patients will continuously be randomized into two groups (Group A and B). Group A will first start the training program and when the training program is finished group B will start the training program. While each group is not performing the training program the patients will be encouraged to physical activity according to their own abilities.
  Results from questionnaires, orthostatic tests and maximal biking tests will be compared between group A and B as well as within each group.
  Interventions: Other: Training program
- Group B - Self-instruction exercise first (Active Comparator): See above.
  Interventions: Other: Training program

INTERVENTIONS:
Other: Training program — A 16-week training program consisting of 2-3 visits per week, and 60 minutes per visit. The program will be done as group exercise under supervision from physiotherapists and/or physicians with special interest in POTS.

SUMMARY:
Postural orthostatic tachycardia syndrome (POTS) is a disorder of unknown origin characterized by orthostatic intolerance and increased heart rate (HR) of ≥ 30 beats/minute during orthostasis in the absence of orthostatic hypotension. In addition to the orthostatic intolerance and tachycardia, patients with POTS experience several debilitating symptoms including light-headedness, nausea, blurred vision, fatigue, mental confusion ("brain-fog"), chest pain and gastrointestinal problems. Several potential underlying mechanisms have been suggested for POTS including autonomic denervation, hypovolemia, hyperadrenergic stimulation and autoantibodies against adrenergic receptors. However, none of these proposed mechanisms has yet led to an effective treatment. Physical activity is recommended as a complimentary treatment in POTS in international guidelines. However, less is known regarding how physical activity could successfully be implemented in clinical practice in patients with POTS. Thus, in the current study, we aim to assess the effect of a 16-week specialized physical activity program in POTS.

DETAILED DESCRIPTION:
A total of 200 patients diagnosed with POTS are asked to participate in the study. The study will be conducted as a cross over study. All POTS patients will continuously be randomized into two groups (Group A and B). Group A will first start the training program and when the training program is finished group B will start the training program. While each group is not performing the training program the patients will be encouraged to physical activity according to their own abilities.

Prior to start of the training program a special POTS questionnaire, the orthostatic hypotension questionnaire and SF-36 (general health questionnaire) will be completed by the participants. Orthostatic tests are performed during 10 minutes, measuring heart rate and blood pressure after 0, 1, 3, and, if possible, 10 minutes of standing. On a separate occasion, patients will perform a maximal biking exercise test, while noting symptoms, degree of exertion, achieved effect, pulse and blood pressure reaction. Following this initial evaluation, the training program will be performed during a total time of 16 weeks, which may be non-consecutive but within 6 months in total. The training program consists of 2-3 visits per week, and 60 minutes per visit. The training may be performed on specialized exercise bicycles in supine position or upright position depending on the severity of POTS symptoms. These exercises will be done under the supervision of physiotherapists with special interest in POTS. After the final training session the POTS questionnaire, the orthostatic hypotension questionnaire and SF-36 will be completed once again. In addition, orthostatic tests and maximal biking exercise test will be performed on a separate occasion soon after the last training session. The POTS questionnaire, the orthostatic hypotension questionnaire, SF-36, hemodynamics and exercise capacity will be compared before and after the 16-weeks training program.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with POTS who have given written informed consent for participation in the study.

Exclusion Criteria:

* Patients with myalgic encephalomyelitis are excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-11-02 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
POTS questionnaire | 12 months
  Subjective symptoms evaluated according to the Malmö POTS Symptom Score which has previously been described (Spahic et al. 2022). The questionnaire is based on patients' own perception of 12 commonly reported symptoms: five cardiac symptoms (palpitations, dizziness, presyncope, dyspnoea and chest pain) and seven non-cardiac symptoms (gastrointestinal symptoms, insomnia, concentration difficulties, headache, myalgia, nausea and fatigue) during the previous 7 days, graded on a scale from 0 (no symptoms) to 10 (very pronounced symptoms). The score ranges from 0 to a maximum score of 120 points.

SECONDARY OUTCOMES:
Orthostatic hypotension questionnaire | 12 months
  Subjective symptoms evaluated according to the orthostatic hypotension questionnaire (OHQ). The OHQ is a questionnaire that has been previously validated and used for orthostatic hypotension but has also been used for quantification of POTS-related symptoms. Further details on the OHQ has previously been described in Kharraziha et al (2020).
SF-36 | 12 months
  Evaluation of 36-item Short Form Health Survey (SF-36). The SF-36 is a 36-item patient-reported questionnaire covering eight health domains: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Orthostatic tests | 12 months
  Hemodynamic measurements (pulse reaction) during orthostatic testing
Maximal biking exercise | 12 months
  Physical capacity measured in watts

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Hamrefors, MD, PhD, Study Director — Department of Clinical Sciences, Lund University; Department of Cardiology Skåne University Hospital
Locations (1):
- Skånes Universitetssjukhus Malmö, Department of Cardiology, Malmo, Sweden

IPD SHARING:
Plan to Share IPD: No
Due to legal and ethical reasons.

REFERENCES:
- [Background] Winker R, Barth A, Bidmon D, Ponocny I, Weber M, Mayr O, Robertson D, Diedrich A, Maier R, Pilger A, Haber P, Rudiger HW. Endurance exercise training in orthostatic intolerance: a randomized, controlled trial. Hypertension. 2005 Mar;45(3):391-8. doi: 10.1161/01.HYP.0000156540.25707.af. Epub 2005 Feb 7. PMID 15699447
- [Background] Fu Q, Vangundy TB, Galbreath MM, Shibata S, Jain M, Hastings JL, Bhella PS, Levine BD. Cardiac origins of the postural orthostatic tachycardia syndrome. J Am Coll Cardiol. 2010 Jun 22;55(25):2858-68. doi: 10.1016/j.jacc.2010.02.043. PMID 20579544
- [Background] George SA, Bivens TB, Howden EJ, Saleem Y, Galbreath MM, Hendrickson D, Fu Q, Levine BD. The international POTS registry: Evaluating the efficacy of an exercise training intervention in a community setting. Heart Rhythm. 2016 Apr;13(4):943-50. doi: 10.1016/j.hrthm.2015.12.012. Epub 2015 Dec 9. PMID 26690066
- [Background] Shibata S, Fu Q, Bivens TB, Hastings JL, Wang W, Levine BD. Short-term exercise training improves the cardiovascular response to exercise in the postural orthostatic tachycardia syndrome. J Physiol. 2012 Aug 1;590(15):3495-505. doi: 10.1113/jphysiol.2012.233858. Epub 2012 May 28. PMID 22641777
- [Background] Kharraziha I, Axelsson J, Ricci F, Di Martino G, Persson M, Sutton R, Fedorowski A, Hamrefors V. Serum Activity Against G Protein-Coupled Receptors and Severity of Orthostatic Symptoms in Postural Orthostatic Tachycardia Syndrome. J Am Heart Assoc. 2020 Aug 4;9(15):e015989. doi: 10.1161/JAHA.120.015989. Epub 2020 Jul 30. PMID 32750291
- [Background] Spahic JM, Hamrefors V, Johansson M, Ricci F, Melander O, Sutton R, Fedorowski A. Malmo POTS symptom score: Assessing symptom burden in postural orthostatic tachycardia syndrome. J Intern Med. 2023 Jan;293(1):91-99. doi: 10.1111/joim.13566. Epub 2022 Sep 16. PMID 36111700
- [Background] Laucis NC, Hays RD, Bhattacharyya T. Scoring the SF-36 in Orthopaedics: A Brief Guide. J Bone Joint Surg Am. 2015 Oct 7;97(19):1628-34. doi: 10.2106/JBJS.O.00030. PMID 26446970
- [Derived] Kharraziha I, Zulj R, Holm H, Fedorowski A, Hamrefors V. Assessing symptom improvement in patients with postural orthostatic tachycardia syndrome (POTS) following a 16-week structured exercise programme: a protocol for a randomised cross-over trial in a clinical outpatient setting. BMJ Open. 2025 Jun 30;15(6):e097057. doi: 10.1136/bmjopen-2024-097057. PMID 40588382